CLINICAL TRIAL: NCT06237686
Title: Clinical Investigation Exploring Two Ostomy Product Prototypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP363
Record Dates: First submitted 2024-01-02; First posted 2024-02-01 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one-armed study (Experimental)
  Interventions: Device: CP363

INTERVENTIONS:
Device: CP363 — All subjects will test both Test product A and B, with a minimum of 7 days apart. In total, each subject will be enrolled in the investigation for 8 days +3 days.

SUMMARY:
Two ostomy product prototypes (Test product A and B) will be tested in this investigation.

All subjects will test both Test product A and B, with a minimum of 7 days apart. In total, each subject will be enrolled in the investigation for 8 days +3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Has given written informed consent
2. Is at least 18 years of age and has full legal capacity
3. Has had an ileostomy for more than 3 months
4. Has suitable peristomal skin area (assessed by investigator)
5. Is currently using flat SenSura Mio 1-piece or 2-piece
6. Has used flat SenSura Mio 1-piece or 2-piece for at least 14 days
7. Has a stoma size less than 45mm in diameter

Exclusion Criteria:

1. Is currently receiving or have within the past 60 days received radio- and/or chemotherapy (Low doses radio- and/or chemotherapy (Assessed by Principal Investigator) is allowed. for indications other than cancer)
2. Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g. lotion or spray or systemic steroid (tablet/injection) treatment
3. Is pregnant or breastfeeding
4. Has dermatological problems in the peristomal area (assessed by investigator)
5. Participates in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol
6. Has any known allergies towards ingredients in the investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One-armed Study
Started (Safety population) | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | One-armed Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 10
Type of stoma [Count of Participants; unit: Participants]
  Ileostomy | 10
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective
Description: Test product A and B's ability to swell around the stoma (assessed by photo/video)
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | One-armed Study
Number analyzed (Participants) | 10
Participants
  Product A. Completely covered in the swelling area | 7
  Product B. Completely covered in the swelling area | 4
  Product A. Partly covered in the swelling area | 1
  Product B. Partly covered in the swelling area | 4
  Product A. Not covered at all in the swelling area | 2
  Product B. Not covered at all in the swelling area | 2
  Product A. Uniform circular swelling | 9
  Product B. Uniform circular swelling | 8
  Product A. No uniform circular swelling | 1
  Product B. No uniform circular swelling | 2

ADVERSE EVENTS:
Time Frame: Each subject was enrolled for 8 days +3 days.
Arm/Group | One-armed Study
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One-armed Study (N=11)
Viral infection (Infections and infestations) | 1 (1) — Not related to the investigational device (Test Product A).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT06237686/Prot_SAP_000.pdf